CLINICAL TRIAL: NCT02104713
Title: A Pilot Safety Study of the Administration of Mesenchymal Stem Cells (MSC) in the Treatment of Burn Wounds
Brief Title: Stem Cell Therapy to Improve Burn Wound Healing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: E.Badiavas (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, E.Badiavas, Professor of Dermatology & Cutaneous Surgery, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20120925
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Skin Burn Degree Second
Keywords: Skin Burn Degree Second; Second degree Burn; Burn wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Allogeneic (MSC's) Application to the Burn Wounds (Experimental): Allogeneic (MSC's) Application to the Burn Wounds. The 1st group of 5 will be started on the lowest dose. If there are no adverse reactions, the 2nd group of 5 will receive a higher dose. This will be repeated for the 3rd and 4th groups with each receiving a higher dose.
  Up to 2 administrations of cells per dose level to be given over a period of no more than 8 weeks. Each administration of cells will be no less than ten days apart and no more than 6 weeks apart.
  Interventions: Biological: Allogeneic (MSC's) Application to the Burn Wounds

INTERVENTIONS:
Biological: Allogeneic (MSC's) Application to the Burn Wounds — Allogeneic (MSC's) Application to the Burn Wounds. The first group of 5 will be started on the lowest dose. If there are no adverse reactions, the second group of 5 will receive a higher dose. This will be repeated for the third and fourth groups with each receiving a higher dose
  1. Initial dose level will be 2.5 x 10³ Allogeneic MSCs cells/square cm.
  2. Second dose level 5 X 10³ Allogeneic MSCs cells/square cm.
  3. Third dose level 1 X 10⁴ Allogeneic MSCs cells/square cm.
  4. Fourth dose level 2 X 10⁴ Allogeneic MSCs cells/square cm.
  Up to 2 administrations of cells will be allowed per dose level to be given over a period of no more than 8 weeks. Each administration of cells will be no less than ten days apart and no more than 6 weeks apart.
  Other Names: Stem Cells Application to the Burn Wounds

SUMMARY:
This study will determine the safety of allogeneic stem cell therapy from healthy donors, for 2nd degree burn wounds of less than 20% Total Body Surface Area (TBSA), at four different dose levels.

Clinical evaluation will take place every 1 to 4 weeks intervals until wound closure, and then monthly for 6 months following the last administration of MSCs.

Once the safety and dose-response analysis in Phase 1 is completed, an expanded trial will be initiated to better examine the efficacy of MSC therapy in 2nd degree burn wounds. Phase 1 will establish the maximum safe dose that will be used in the Phase II trial.

ELIGIBILITY:
- Donors:

Eligibility Criteria:

* No history of malignancy
* No active coagulopathy and/or hypocoagulable state
* No history of cardio/pulmonary conditions
* Negative tests for Hepatitis A, Hepatitis B, Hepatitis C, RPR, HIV 1 / 2, HTLV I/II, Chagas Disease, NAT for HCV, HIV and WNV.
* Hemoglobin ≥ 13.0 g/dL
* Platelet count 140,000 to 440,000/ul
* WBC 3.0 to 11.0 K/ul
* BNP ≤ 100 pg /mL
* No anomalies on the CBC and differential suggestive of a hematopoietic disorder
* Creatinine ≤ 1.5 mg/dL
* ALT ≤ 112 IU/L
* AST ≤ 100 IU/L
* Bilirubin < 1.5 mg/dL
* No diabetes
* Systolic blood pressure ≤ 170
* Diastolic blood pressure ≤ 90
* No history of autoimmune disorders

Recipients:

Inclusion Criteria:

1. Male or female subjects 18 years of age or older with Superficial, Intermediate or Deep 2nd Degree Burn Wounds
2. Injury within the prior 7 days
3. Subjects must understand and give written informed consent.
4. Subjects must agree to have biopsies performed as per protocol
5. Subjects must be accessible for weekly wound treatment and assessment visits
6. Males and females must agree to use an acceptable method of contraception. Exceptions will be females of non-childbearing age and monogamous males who are partners of females of non-childbearing age. Acceptable methods of birth control include; history of sterilization, birth control pills, depoprogesterone injections, a barrier contraceptive such as a condom with or without spermicide cream or gel, diaphragms or cervical cap with or without spermicide cream or gel, or an intrauterine device (IUD).
7. Maximum wound size limited to:

   * Single wound: ≤ 5% body surface area (BSA)
   * Multiple wounds treated in a defined anatomical region with ≤ 20% cumulative BSA.
8. Diabetic subjects: HbA1c ≤ 8%

Exclusion Criteria:

1. Solely 1st degree or solely 3rd degree burns
2. Subjects with superficial 2nd degree burn who are expected to heal within 2 weeks post standard therapy
3. Evidence of active infection at the wound site
4. Evidence of significant wound healing prior to treatment
5. Wound located in the area of fingers, toes, face, or perineum
6. Wound where 75% or more extends across joints
7. Electrical or chemical burns
8. Have any requirement for the use of systemic steroids or immunosuppressive
9. Subjects Allergic to human albumin, streptomycin, or penicillin
10. Be a pregnant female or nursing mother
11. Subjects who are known or found to be HIV positive
12. Current history of alcohol or substance abuse or history of alcohol or substance abuse requiring treatment within the past 12 months
13. Patients with severe medical conditions

    1. Malignancy (other than non melanoma skin cancer) not in remission or in remission less than 5 years
    2. Life expectancy less than two years
    3. Severe cardiopulmonary disease restricting ambulation to the clinical facility
14. WBC <3 or > 10 x10⁹/L, Hgb < 9g/dL, platelets count 100x10⁹/L or less, serum creatinine > 1.5 times the upper normal limit, AST or ALT > 2.5 times the upper normal limit.
15. Subjects with abnormal bilirubin levels.
16. Subjects with abnormal PT/INR laboratory values while not on chronic anticoagulant treatment which can be held for minor surgical procedures
17. Those with a known history of coagulopathy
18. Subjects who are potential recipients of tissue or organ transplantation
19. Subjects with circulating Hepatitis B antigen and/or who are seropositive for Hepatitis C antibody
20. History of poor compliance, unreliability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Monitoring for adverse events as Assessed by CTCAE v4.0 following administration of allogeneic MSCs to 2nd degree burn wounds. | 1.5 years
  The study will consist of a dose escalation phase consisting of four dose levels. Each dose level will compare the safety of administering allogeneic MSCs, with 5 patients per group.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Schulman, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maranda EL, Wang MX, Shareef S, Tompkins BA, Emerson C, Badiavas EV. Surgical management of leukoderma after burn: A review. Burns. 2018 Mar;44(2):256-262. doi: 10.1016/j.burns.2017.05.004. Epub 2017 Jun 8. PMID 28602587